CLINICAL TRIAL: NCT04073433
Title: A Phase 1, Open-Label, Multi-Site Study to Assess Psychological Effects of MDMA-Assisted Psychotherapy When Administered to Healthy Volunteers
Brief Title: Psychological Effects of Methylenedioxymethamphetamine (MDMA) When Administered to Healthy Volunteers (MT-2)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MT2
Record Dates: First submitted 2019-07-30; First posted 2019-08-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Psychological Effects of Study Drug
Keywords: Mood; Subjective Effects; MDMA
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDMA-assisted therapy (Experimental): One session of MDMA-assisted therapy with a dose of 120 mg midomafetamine HCl and optional supplemental dose of 60 mg 1.5 to 2 hours later
  Interventions: Drug: Midomafetamine HCl; Behavioral: Therapy

INTERVENTIONS:
Drug: Midomafetamine HCl — 120 mg midomafetamine HCl
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA; midomafetamine; MDMA HCl
Behavioral: Therapy — Non-directive therapy conducted during MDMA-assisted therapy session

SUMMARY:
The goal of this clinical trial is to study MDMA-assisted therapy in healthy volunteers and provide training of therapists. The main question it aims to answer is:

Does MDMA-assisted therapy result in personal and professional benefits?

Participants will have a non-drug preparatory session prior to each experimental session and an integrative session after each experimental session.

DETAILED DESCRIPTION:
The Phase 1, randomized, placebo-controlled study MT1 was designed to collect safety and quantitative data on mood, psychological symptoms, personality traits, and interpersonal closeness in therapists learning to conduct MDMA-assisted psychotherapy or MDMA research among 120 healthy volunteers. The MT1 study was also designed to expand the knowledge of therapists training to conduct MDMA-assisted psychotherapy research. In the MT1 study, several participants submitted optional written narratives with impressions that participating in MDMA-assisted psychotherapy helped them professionally and personally.

This Phase 1, open-label, multi-site research study is designed to build upon the MT1 study to further assess the psychological effects and safety of manualized MDMA-assisted psychotherapy, while supporting the expansion of knowledge for treatment providers who are learning to conduct MDMA-assisted psychotherapy or MDMA research. This study is intended to look further into the personal and professional benefits spontaneously reported in narratives to the site team from the MT1 study participants. This will be done by collecting changes in self-compassion, burnout, professional quality of life, psychological inflexibility, and mood using validated measures in a larger sample of treatment providers, allowing for effect size calculations.

ELIGIBILITY:
Inclusion Criteria:

* Are learning to conduct MDMA-assisted psychotherapy or MDMA research through the MDMA Therapy Training Program
* Are at least 18 years old
* Are fluent in speaking and reading the predominantly used or recognized language of the study site
* Are able to swallow pills
* Must provide a contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the investigator in the event of an emergency or if the participant is unreachable
* Must agree to inform the investigators within 48 hours if any medical conditions occur or medical procedures are planned
* If of childbearing potential, must have a negative pregnancy test at study entry and prior to the Experimental Session, and must agree to use adequate birth control through 10 days after the Experimental Session
* If nursing, must be willing to dispose of breastmilk from dosing through 5 days after each Experimental Session
* Must not participate in any other interventional clinical trials during the duration of the study
* Must agree to not operate a vehicle for at least 24 hours after initial drug administration.
* Must have transportation available after the Experimental Session and through the following day, for traveling back for the Integrative Session.
* Must commit to medication dosing, therapy, and study procedures
* Are willing to be contacted via telephone for all necessary telephone contacts.

Exclusion Criteria:

* Are not able to give adequate informed consent
* Have uncontrolled hypertension
* Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] in males and >460 ms in females corrected by Bazett's formula)
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Have evidence or history of significant medical disorders
* Have symptomatic liver disease
* Have history of hyponatremia or hyperthermia
* Weigh less than 45 kilograms (kg)
* Are pregnant, or are of childbearing potential and are not practicing an effective means of birth control
* Have any current problematic patterns of alcohol or other substance use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Self Compassion Scale (SCS) total score | 9 weeks post-enrollment
  Self Compassion Scale (SCS) total score, a 26-item self-report measure of self-compassion

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Ot'alora, Principal Investigator — Private Practice